CLINICAL TRIAL: NCT02960724
Title: Phase II Trial: uPAR PET/CT for Staging Advanced and Localised Oral and Oropharyngeal Cancer
Brief Title: uPAR PET/CT for Staging Advanced and Localised Oral and Oropharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kirstine Karnov, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK-2016-HHC1
Record Dates: First submitted 2016-10-11; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Oral Cancer; Oropharyngeal Cancer; Neoplasms; Head and Neck Neoplasms; Cancer of Mouth; Neoplasms by Site
Keywords: Uroplasminogen Plasminogen Activator Receptor; Oropharyngeal cancer; oral cancer; Positron Emission Tomography
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Neoplasms; Head and Neck Neoplasms; Neoplasms by Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-AE105 PET/CT (Experimental): One injection of 68Ga-NOTA-AE105 followed by positron emission tomography/computed tomography (PET/CT scan) will be performed before surgery and compared with the histological findings to evaluate uPAR PET/CT in staging of oral cancer and oropharyngeal cancer.
  Interventions: Other: 68Ga-NOTA-AE105 PET/CT

INTERVENTIONS:
Other: 68Ga-NOTA-AE105 PET/CT — One injection of 68Ga-NOTA-AE105 (app. 200 Mbq) followed by Positron Emission Tomography Scan.

SUMMARY:
uPAR PET/CT for Staging Advanced and Localised oral and oropharyngeal cancer

DETAILED DESCRIPTION:
To compare the diagnostic value of uPAR-PET/CT for prognostication compared to the current imaging options (CT, MRI and ultrasound) by observer-blinded readings. The reference that will be used as "gold standard" is the pathological examination of the surgically removed tissues.

The new imaging modality (uPAR-PET/CT) will be used in two separate groups of patients with head and neck cancer:

Study I:

Patients with oral cancer without clinical evidence of spread (OSCC in stage cN0)

Study II:

Patients with metastatic oral cancer (OSCC in stage cN +) and patients with metastatic oropharyngeal cancer (OPSCC in stage cN +).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand patient information and to give informed consent
* Not previously irradiated or operated on neck
* Operable disease

Study I OSCC cN0 verified histologically by pathologic examination of biopsy

Study II OSCC or OPSCC N + verified histologically by pathologic examination of biopsy

Exclusion Criteria:

* Pregnancy
* Patients who are candidates for curative intentional radiation
* Patients who have had surgery or radiation therapy to the neck as this may alter the lymph drainage.
* Other diseases assessed by the investigator as basis for exclusion.
* Age under 18 or over 85 years
* Obesity> 140 kg
* Allergy to 68Ga-NOTA-AE105

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The number of lymph node metastases that can be identified by means of uPAR PET / CT compared with the histological findings. | Through study completion, an average of 1.5 year

SECONDARY OUTCOMES:
Evaluation of the correlation between uPAR PET signal (quantified as SUVmax) and the immunohistochemical expression of uPAR evaluated by an H-score (intensity x the percentage of stained tumor tissues throughout the tumor margin). | Through study completion, an average of 1.5 year
Evaluation of the correlation between tumor burden (assessed v.h.a. TNM staging) uPAR-PET signal (assessed as SUVmax) and the amount of uPAR metabolites in plasma. | Through study completion, an average of 1.5 year
Determination of the lower detection limit of the amount of tumor tissue for uPAR-PET correlated with the histological H-score x tumor size (where tumor size is evaluated on the pathological preparation of pathologist) | Through study completion, an average of 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, MD,DMSc,PhD, Study Director — Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Skovgaard D, Persson M, Brandt-Larsen M, Christensen C, Madsen J, Klausen TL, Holm S, Andersen FL, Loft A, Berthelsen AK, Pappot H, Brasso K, Kroman N, Hojgaard L, Kjaer A. Safety, Dosimetry, and Tumor Detection Ability of 68Ga-NOTA-AE105: First-in-Human Study of a Novel Radioligand for uPAR PET Imaging. J Nucl Med. 2017 Mar;58(3):379-386. doi: 10.2967/jnumed.116.178970. Epub 2016 Sep 8. PMID 27609788
- [Result] Persson M, Skovgaard D, Brandt-Larsen M, Christensen C, Madsen J, Nielsen CH, Thurison T, Klausen TL, Holm S, Loft A, Berthelsen AK, Ploug M, Pappot H, Brasso K, Kroman N, Hojgaard L, Kjaer A. First-in-human uPAR PET: Imaging of Cancer Aggressiveness. Theranostics. 2015 Sep 13;5(12):1303-16. doi: 10.7150/thno.12956. eCollection 2015. PMID 26516369
- [Result] Persson M, Nedergaard MK, Brandt-Larsen M, Skovgaard D, Jorgensen JT, Michaelsen SR, Madsen J, Lassen U, Poulsen HS, Kjaer A. Urokinase-Type Plasminogen Activator Receptor as a Potential PET Biomarker in Glioblastoma. J Nucl Med. 2016 Feb;57(2):272-8. doi: 10.2967/jnumed.115.161703. Epub 2015 Oct 1. PMID 26429955